CLINICAL TRIAL: NCT06569615
Title: Efficacy of Extracorporeal Shock Wave Therapy, LASER Therapy and Cryotherapy on PPT, Pain and Functional Disability in Patients Having Sacroiliitis: A Randomized Control Study
Brief Title: Efficacy of Extracorporeal Shock Wave Therapy, LASER Therapy and Cryotherapy in Patients Having Sacroiliitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Najran University (Other)
Responsible Party: Principal Investigator, Hashim Ahmed, Assistant Professor, Najran University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202406-076-021198-048523
Record Dates: First submitted 2024-08-19; First posted 2024-08-26 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Sacroilitis
MeSH Terms: interventions — Extracorporeal Shockwave Therapy; Laser Therapy; Cryotherapy; Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): shock wave Group
  Interventions: Other: shock wave therapy; Other: Exercises
- Group 2 (Experimental): LASER Group
  Interventions: Other: LASER Therapy; Other: Exercises
- Group 3 (Experimental): Cryotherapy Group
  Interventions: Other: Cryotherapy; Other: Exercises

INTERVENTIONS:
Other: shock wave therapy — All the participants in first week will receive the ice pack for 15 minutes 3 times a day at the lumbosacral area to reduce inflammation in the area, along with rest to reduce irritation at the lumbosacral area for the first week.
  From the 2nd week:
  Participants will be given Radial shockwave therapy, (Storz Medical Shock Master MP200 device) for 10 minutes/session, one session/week, for 8 weeks.
  Arms: Group 1
Other: LASER Therapy — All the participants in first week will receive the ice pack for 15 minutes 3 times a day at the lumbosacral area to reduce inflammation in the area, along with rest to reduce irritation at the lumbosacral area for the first week.
  From the 2nd week:
  Participants will be given LASER, (LEVELASER EZ1 EASYONE) over the lumbosacral area for 10 minutes/Session, three session/week, for 8 weeks.
  Arms: Group 2
Other: Cryotherapy — All the participants in first week will receive the ice pack for 15 minutes 3 times a day at the lumbosacral area to reduce inflammation in the area, along with rest to reduce irritation at the lumbosacral area for the first week.
  From the 2nd week:
  Participants will be given Cryotherapy, (Gymna UniphyCryoflow 1000 IR Shock Master ICE-CT device) over the lumbosacral area for 10 minutes/Session, three session/week, for 8 weeks.
  Arms: Group 3
Other: Exercises — The assigned exercises for all participants will include 1. Bilateral bridging, 2. Knee to chest, 3. Back extension within a pain-free range, 4. Plank, 5. Baby pose stretch, 6. Cat and camel, 7. Bilateral adductor ball squeezes and 8. Stretching exercise (Gluteal /Piriformis stretch, Quads /Hams stretch. The treatment plan involved performing three sets of exercises, with each set comprising 8 to 10 repetitions. 20-30 minutes of exercise session will be conducted three times per week over a span of 8 weeks.

SUMMARY:
This research aimed to determine the effect of extracorporeal shock wave therapy, LASER therapy and cryotherapy on PPT, Pain and functional disability in patients having Sacroiliitis.

DETAILED DESCRIPTION:
The study will be based on a three-arm parallel group randomized control design. sixty participants of sacroiliitis will be recruited from the Physiotherapy department, at Najran University, K.S.A. Study objectives and procedure will be properly explained and written informed consent will be obtained at the beginning of the study. All the participants will be randomly divided into three groups 1, 2 and 3.

All the participants in first week will receive the ice pack for 15 minutes 3 times a day at the lumbosacral area to reduce inflammation in the area, along with rest to reduce irritation at the lumbosacral area for the first week.

From the 2nd week:

Group 1 will be administered ESWT plus exercise, Group 2 will be administered LASER plus exercise, and Group 3 will be administered cryotherapy and exercise.

ELIGIBILITY:
Inclusion Criteria:

* Pain in one or both buttocks, hip pain, thigh pain, or even pain more distal.
* Patients may report that their pain is worse after sitting for prolonged periods or with rotational movements that will be intensified when bending laterally or backward and
* Positive outcome in a minimum of three out of five pain-provocation tests (i.e., compression test, distraction test, Faber sign, Gaenslen test, and thigh thrust.
* Pain close to the posterior superior iliac spine and the patient could point with a single finger to the location of pain (Fortin Finger Test).

Exclusion Criteria:

* The Participant who had undergone surgery or experienced significant trauma to the spine, pelvis, lower limb, chest, or abdomen within the past 12 months.
* The participants with lower extremity musculoskeletal disorders, localized spinal pathology, congenital anomalies of the hip, pelvis, or spine that limited mobility.
* having a positive straight leg raising test
* receiving nonsteroidal anti-inflammatory drugs, hormonal therapy, or corticosteroid injections
* individuals with tumors, fractures. ankylosing spondylitis.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-09-25 (Estimated)

PRIMARY OUTCOMES:
Pain Pressure Threshold (PPT) | 8 Weeks
  Pain pressure threshold of muscle tenderness will be measured by using the algometer
Pain Intensity | 8 Weeks
  Pain intensity will be measured by using the Visual Analogue Scale (VAS),a linear scale wherein patients indicate their pain intensity on a 10 cm line ranging from 'no pain' to 'worst imaginable pain'

SECONDARY OUTCOMES:
Functional Disability | 8 Weeks
  Functional disability will be measured by using the Oswestry Disability Index (ODI),a validated 10-item questionnaire evaluating various dimensions of daily living

CONTACTS AND LOCATIONS:
Overall Officials: Hashim Ahmed, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Hashim Ahmed, Najrān, Najran Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No